CLINICAL TRIAL: NCT03247517
Title: Evaluation of SPN 812 (Viloxazine Extended-release Capsule) 200 and 400 mg Efficacy and Safety in Adolescents With ADHD - A Double-Blind, Placebo-Controlled, Pivotal Trial
Brief Title: Evaluation of SPN-812 (Viloxazine Extended-release Capsule) Low Dose in Adolescents With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 812P302
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo, qd, oral capsule
  Interventions: Drug: Placebo
- 200mg SPN-812 (Experimental): 200mg SPN-812, qd, oral capsule
  Interventions: Drug: 200mg SPN-812
- 400mg SPN-812 (Experimental): 400mg SPN-812, qd, oral capsule
  Interventions: Drug: 400mg SPN-812

INTERVENTIONS:
Drug: Placebo — Placebo was administered once daily
  Other Names: PBO
  Arms: Placebo
Drug: 200mg SPN-812 — 200mg SPN-812 was administered once daily and compared to placebo
  Other Names: SPN-812
  Arms: 200mg SPN-812
Drug: 400mg SPN-812 — 400mg SPN-812 was administered once daily and compared to placebo
  Other Names: SPN-812
  Arms: 400mg SPN-812

SUMMARY:
This study will evaluate the efficacy and safety of low doses of SPN-812 in adolescents 12-17 years of age.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, 3-arm, parallel-group study, to assess the efficacy and safety of SPN-812 as monotherapy for the treatment of adolescents 12-17 years old with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects, 12-17 years of age, inclusive.
2. Diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5), confirmed with the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
3. Attention Deficit/Hyperactivity Disorder Rating Scale-5-Home Version: Adolescent, Investigator Administered and Scored (ADHD-RS-5) score of at least 28.
4. CGI-S score of at least 4 at screening.
5. Weight of at least 35 kg.
6. Free of medication for the treatment of ADHD for at least one week prior to randomization and agreement to remain so throughout the study.
7. Considered medically healthy by the Investigator via assessment of physical examination, medical history, clinical laboratory tests, vital signs, and electrocardiogram.
8. Written informed consent obtained from the subject's parent or legal representative and informed assent from the subject, if applicable.
9. Females of childbearing potential (FOCP) must be either sexually inactive (abstinent) or, if sexually active, must agree to use one of the following acceptable birth control methods beginning 30 days prior to the first dose, throughout the study:

   1. simultaneous use of male condom and intra-uterine contraceptive device placed at least four weeks prior to the first study drug administration
   2. surgically sterile male partner
   3. simultaneous use of male condom and diaphragm with spermicide
   4. established hormonal contraceptive

Exclusion Criteria:

1. Current diagnosis of major psychiatric disorders. Subjects with Major Depressive Disorder are allowed in the study if the subject is free of episodes both currently and for the last six months.
2. Current diagnosis of major neurological disorders. Subjects with seizures or a history of seizure disorder within the immediate family (siblings, parents), or a history of seizure-like events are excluded from the study.
3. Current diagnosis of significant systemic disease.
4. Evidence of suicidality (defined as either active suicidal plan/intent or active suicidal thoughts, or more than one lifetime suicide attempt) within the six months before Screening or at Screening.
5. BMI greater than 95th percentile for the appropriate age and gender.
6. History of an allergic reaction to viloxazine or related drugs.
7. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Investigator, could contraindicate the subject's participation in this study.
8. Subjects who received any investigational drug within the longer of 30 days or 5 half-lives prior to Day 1 dosing of SM.
9. Any reason, which, in the opinion of the Investigator, would prevent the subject from participating in the study
10. Positive screen for drugs of abuse at the Screening Visit. A positive test for amphetamines is allowed for subjects receiving a stimulant ADHD medication at Screening as long as the subject agrees to discontinue the stimulant for the duration of the study beginning at least one week prior to the Baseline Visit.
11. Pregnancy or refusal to practice abstinence or acceptable birth control during the study (for female subjects of childbearing potential)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schwabe, Study Director — Supernus Pharmaceuticals, Inc.
Locations (12):
- United States (12):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Miami Clinical Research, Miami, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Texas Physicians Medical Research Group, Arlington, Texas
  - Houston Clinical Trials, Houston, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faraone SV, Gomeni R, Hull JT, Busse GD, Lujan B, Rubin J, Nasser A. Response of peer relations and social activities to treatment with viloxazine extended-release capsules (Qelbree(R) ): A post hoc analysis of four randomized clinical trials of children and adolescents with attention-deficit/hyperactivity disorder. Brain Behav. 2023 Apr;13(4):e2910. doi: 10.1002/brb3.2910. Epub 2023 Feb 27. PMID 36847750
- [Derived] Faraone SV, Gomeni R, Hull JT, Busse GD, Melyan Z, Rubin J, Nasser A. Executive Function Outcome of Treatment with Viloxazine Extended-Release Capsules in Children and Adolescents with Attention-Deficit/Hyperactivity Disorder: A Post-Hoc Analysis of Four Randomized Clinical Trials. Paediatr Drugs. 2021 Nov;23(6):583-589. doi: 10.1007/s40272-021-00470-2. Epub 2021 Sep 15. PMID 34523063
- [Derived] Nasser A, Kosheleff AR, Hull JT, Liranso T, Qin P, Busse GD, Fava M, Maletic V, Rubin J, Lopez F. Evaluating the likelihood to be helped or harmed after treatment with viloxazine extended-release in children and adolescents with attention-deficit/hyperactivity disorder. Int J Clin Pract. 2021 Aug;75(8):e14330. doi: 10.1111/ijcp.14330. Epub 2021 May 26. PMID 33971070
- [Derived] Nasser A, Kosheleff AR, Hull JT, Liranso T, Qin P, Busse GD, O'Neal W, Fava M, Faraone SV, Rubin J. Translating Attention-Deficit/Hyperactivity Disorder Rating Scale-5 and Weiss Functional Impairment Rating Scale-Parent Effectiveness Scores into Clinical Global Impressions Clinical Significance Levels in Four Randomized Clinical Trials of SPN-812 (Viloxazine Extended-Release) in Children and Adolescents with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2021 Apr;31(3):214-226. doi: 10.1089/cap.2020.0148. Epub 2021 Feb 17. PMID 33600233

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo oral capsule
  Treatment A: Placebo will be administered once daily
- 200mg SPN-812: 200mg SPN-812 oral capsule
  Treatment B: SPN-812 was administered once daily and compared to placebo
- 400mg SPN-812: 400mg SPN-812 oral capsule
  Treatment C: SPN-812 was administered once daily and compared to placebo
Period: Overall Study
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
Started (The number of subjects reported here is based on the Safety Population (assigned treatment arm); includes subjects who were randomized and took at least one dose of study medication.) | 104 | 98 | 106 (One subject randomized to the 400mg/day SPN-812 arm received 200mg/day SPN-812 during the trial)
Completed | 96 | 78 | 92
Not Completed | 8 | 20 | 14
Not completed — Adverse Event | 0 | 4 | 2
Not completed — Lost to Follow-up | 2 | 6 | 4
Not completed — Consent withdrawn by caregiver | 1 | 4 | 7
Not completed — Assent/consent withdrawn by subject | 2 | 3 | 1
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Multiple reasons | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: The ITT population includes subjects who were randomized, took at least one dose of study medication, have a baseline Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) assessment and have at least one post-baseline ADHD-RS-5 assessment.
Groups:
- 200mg SPN-812: 200mg SPN-812 oral capsule
  Treatment B: SPN-812 will be administered once daily and compared to placebo
- 400mg SPN-812: 400mg SPN-812 oral capsule
  Treatment C: SPN-812 will be administered once daily and compared to placebo
- Total: Total of all reporting groups
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812 | Total
Number analyzed (Participants) | 104 | 94 | 103 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.60) | 13.9 (1.48) | 14.0 (1.59) | 13.9 (1.56)
Age, Customized [Count of Participants; unit: Participants]
  12 to 14 years | 70 | 63 | 64 | 197
  15 to 17 years | 34 | 31 | 39 | 104
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 28 | 36 | 110
  Male | 58 | 66 | 67 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 27 | 32 | 89
  Not Hispanic or Latino | 74 | 67 | 71 | 212
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 3
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 39 | 37 | 42 | 118
  White | 63 | 53 | 55 | 171
  More than one race | 2 | 2 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 104 | 94 | 103 | 301
ADHD-RS-5 Total Score [Mean (Standard Deviation); unit: units on a scale] — The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. It consists of 18 items that correspond to the 18 ADHD symptoms per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). Each item is rated on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). Total score = sum of 18 items (range: 0 to 54). The higher the score, the more severe the ADHD symptoms (a total score >=28 was an inclusion criterion of this study).
  units on a scale | 40.5 (6.79) | 39.9 (7.22) | 39.4 (7.59) | 39.9 (7.20)
ADHD-RS-5 Inattention [Mean (Standard Deviation); unit: units on a scale] — The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. It consists of 18 items that correspond to 18 ADHD symptoms per DSM-5, including 9 items for the Hyperactivity/Impulsivity (HI) subscale and 9 items for the Inattention (IA) subscale. Each item is rated on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). The IA Subscale score = sum of all 9 IA items on the ADHD-RS-5 (range: 0 to 27). The higher the score, the more severe the IA symptoms of ADHD.
  units on a scale | 22.4 (3.67) | 22.2 (3.66) | 21.5 (3.60) | 22.0 (3.65)
ADHD-RS-5 Hyperactivity/Impulsivity [Mean (Standard Deviation); unit: units on a scale] — The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. It consists of 18 items that correspond to 18 ADHD symptoms per DSM-5, including 9 items for the Hyperactivity/Impulsivity (HI) subscale and 9 items for the Inattention (IA) subscale. Each item is rated on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). The HI Subscale score = sum of all 9 HI items on the ADHD-RS-5 (range: 0 to 27). The higher the score, the more severe the HI symptoms of ADHD.
  units on a scale | 18.1 (5.35) | 17.7 (5.71) | 17.9 (5.64) | 17.9 (5.55)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of SPN-812 Assessed by Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5)
Description: The Primary Endpoint was the change from baseline in the Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) Total score at Week 6 (End of Study). The ADHD-RS-5 is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) symptoms of ADHD. Each item is rated on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). A Total score is calculated by adding the responses of all 18 items (range: 0-54; the higher the score, the more severe the ADHD symptoms). Lower change from baseline scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo oral capsule
  Treatment A: Placebo was administered once daily
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 104 | 94 | 103
units on a scale | -11.4 (1.37) | -16.0 (1.45) | -16.5 (1.38)
Statistical Analysis 1: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.0232, Mixed Models for Repeated Measures; Least Square Mean Difference = -4.5, 95% CI 2-sided [-8.4 to -0.6], Standard Error of Mean 1.98
Statistical Analysis 2: Comparison: Placebo vs 400mg SPN-812; Test type: Superiority; p = 0.0091, Mixed Models for Repeated Measures; Least Square Mean Difference = -5.1, 95% CI 2-sided [-8.9 to -1.3], Standard Error of Mean 1.93

2. Secondary Outcome: Effect of SPN-812 Assessed by Clinical Global Impression-Improvement (CGI-I) Scale
Description: The first Key Secondary Endpoint was the Clinical Global Impression-Improvement (CGI-I) Scale score at Week 6 (End of Study). The CGI-I scale is a single item assessment of how much the patient's illness has improved or worsened relative to a baseline state prior to the beginning of treatment. The CGI-I is rated on a 7-point Likert scale from 1 to 7, where 1 = "very much improved" and 7 = "very much worse." Successful therapy is indicated by a lower overall score in subsequent testing.
Time Frame: Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 104 | 94 | 103
units on a scale | 3.0 (0.11) | 2.5 (0.12) | 2.4 (0.12)
Statistical Analysis 1: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.0042, ANCOVA; ANCOVA model with baseline Clinical Global Impression-Severity of Illness (CGI-S) score and treatment as fixed independent variables; Least Square Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Placebo vs 400mg SPN-812; Test type: Superiority; p = 0.0003, ANCOVA; [statistical method as in outcome 2, analysis 1]; Least Square Mean Difference = -0.6, 95% CI 2-sided [-0.9 to -0.3], Standard Error of Mean 0.16

3. Secondary Outcome: Effect of SPN-812 Assessed by Conners 3rd Edition - Parent Short Form (C3-PS)
Description: The second Key Secondary Endpoint was the change from baseline in the Conners 3rd Edition - Parent Short Form (C3PS) Composite T-score at Week 6 (End of Study). The Conners 3rd Edition is a focused diagnostic tool for the assessment of ADHD and associated learning, behavior, and emotional problems in children 6 to 18 years of age. The C3PS is completed by a child's parent/guardian and is comprised of 45 items with subsets of items related to six content scales: inattention, hyperactivity/impulsivity, executive functioning, learning problems, defiance/aggression and peer relations. The parent rates his/her child on the first 43 items of the C3PS using a 4-point Likert scale (0-3; where 0=not at all true [never, seldom] and 3=very much true [very often, very frequently]) based on past month; the last 2 items are fill-in-the-blank and do not contribute to the raw score(s). Raw scores are converted to T-scores. Lower change from baseline T-scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 104 | 94 | 103
T-score | -5.7 (1.04) | -6.4 (1.12) | -8.6 (1.07)
Statistical Analysis 1: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.6854, ANCOVA; Least Square Mean Difference = -0.6, 95% CI 2-sided [-3.6 to 2.4], Standard Error of Mean 1.54
Statistical Analysis 2: Comparison: Placebo vs 400mg SPN-812; Test type: Superiority; p = 0.0518, ANCOVA; Least Square Mean Difference = -2.9, 95% CI 2-sided [-5.8 to 0.0], Standard Error of Mean 1.49

4. Secondary Outcome: Effect of SPN-812 Assessed by Weiss Functional Impairment Rating Scale-Parent Report (WFIRS-P)
Description: The third Key Secondary Endpoint was the change from baseline in the Weiss Functional Impairment Rating Scale-Parent Report (WFIRS-P) Total Average score at Week 6 (End of Study). The WFIRS instrument evaluates ADHD-related functional impairment. The WFIRS-P is completed by the child's parent/guardian and is comprised of 50 items grouped into six domains: Family (10 items), School (10 items, includes learning [4 items] and behavior [6 items]), Life Skills (10 items), Child's Self-Concept (3 items), Social Activities (7 items), and Risky Activities (10 items). The parent/guardian rates each item on a 4-point Likert scale (0-3; where 0=never or not at all to 3= very often or very much) based on their child's behavior past month. A Total Average score was computed by calculating mean rating of all 50 items (ranging from 0 to 3, where a higher value represents more severe functional impairment). Lower change from baseline Total Average scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 104 | 94 | 103
units on a scale | -0.19 (0.041) | -0.27 (0.045) | -0.31 (0.042)
Statistical Analysis 1: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.2062, ANCOVA; Least Square Mean Difference = -0.08, 95% CI 2-sided [-0.20 to 0.04], Standard Error of Mean 0.061
Statistical Analysis 2: Comparison: Placebo vs 400mg SPN-812; Test type: Superiority; p = 0.0519, ANCOVA; Least Square Mean Difference = -0.11, 95% CI 2-sided [-0.23 to 0.00], Standard Error of Mean 0.059

5. Secondary Outcome: Effect of SPN-812 Assessed by 50% Responder Rate Per the Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5)
Description: An additional secondary endpoint was the percentage of responders at Week 6 (End of Study). A responder was defined as a subject who had a 50% or greater reduction (improvement) in their change from baseline Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) Total score at Week 6 (End of Study). Values range from 0 to 100%. A higher percentage represents a greater number of responders.
Time Frame: Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 104 | 94 | 103
percentage of subjects | 27.0 | 45.8 | 44.6
Statistical Analysis 1: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.0068, Regression, Logistic; Risk Difference (RD) = 18.8, 95% CI 2-sided [5.5 to 32.2]
Statistical Analysis 2: Comparison: Placebo vs 400mg SPN-812; Test type: Superiority; p = 0.0095, Regression, Logistic; Risk Difference (RD) = 17.6, 95% CI 2-sided [4.6 to 30.5]

6. Secondary Outcome: Effect of SPN-812 Assessed by Stress Index for Parents of Adolescents (SIPA)
Description: Another secondary endpoint was the change from baseline in the Stress Index for Parents of Adolescents (SIPA) Total score to Week 6 (End of Study). The SIPA is a 112-item screening/diagnostic instrument for parents of adolescents 11-19 years of age that identifies areas of stress in parent-adolescent interactions. Items 1-90 are rated on a 5-point Likert scale (where SD=Strongly Disagree, D=Disagree, NS=Not Sure, A=Agree, and SA=Strongly Agree) and yields a raw score for 3 Domains (Adolescent Domain, Parent Domain, and Adolescent-Parent Domain) that focus on a parent's perception of their child's personality and on the parent's characteristics and behaviors. The sum of the 3 Domain scores yields the Total (Parent Stress) score (range: 90-450; higher total scores indicate higher levels of stress). Lower change from baseline scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 104 | 94 | 103
units on a scale | -13.7 (3.72) | -12.0 (4.08) | -15.3 (3.83)
Statistical Analysis 1: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.7629, ANCOVA; Least Square Mean Difference = 1.7, 95% CI 2-sided [-9.1 to 12.5], Standard Error of Mean 5.51
Statistical Analysis 2: Comparison: Placebo vs 400mg SPN-812; Test type: Superiority; p = 0.7648, ANCOVA; Least Square Mean Difference = -1.6, 95% CI 2-sided [-12.1 to 8.9], Standard Error of Mean 5.36

7. Secondary Outcome: Effect of SPN-812 Assessed by the Hyperactivity/Impulsivity Subscale and the Inattention Subscale of the Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5)
Description: An additional secondary endpoint was the change from baseline in the Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) Hyperactivity/Impulsivity subscale score and Inattention subscale score at Week 6 (End of Study). The ADHD-RS-5 is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 DSM-5 symptoms of ADHD, including 9 items for the Hyperactivity/Impulsivity subscale and 9 items for the Inattention subscale. Each item is rated on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). Each subscale score is calculated by adding the responses of all respective 9 items (range: 0-27; the higher the subscale score, the more severe the Hyperactivity/Impulsivity or Inattention symptoms). Lower change from baseline subscale scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 104 | 94 | 103
units on a scale
  Hyperactivity/Impulsivity subscale | -5.1 (0.69) | -7.7 (0.73) | -8.4 (0.69)
  Inattention subscale | -6.6 (0.74) | -8.7 (0.78) | -8.7 (0.74)
Statistical Analysis 1: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to the Hyperactivity/Impulsivity subscale score; Test type: Superiority; p = 0.0069, ANCOVA; Least Square Mean Difference = -2.7, 95% CI 2-sided [-4.6 to -0.7], Standard Error of Mean 0.99
Statistical Analysis 2: Comparison: Placebo vs 400mg SPN-812; This analysis pertains to the Hyperactivity/Impulsivity subscale score; Test type: Superiority; p = 0.0005, ANCOVA; Least Square Mean Difference = -3.4, 95% CI 2-sided [-5.2 to -1.5], Standard Error of Mean 0.96
Statistical Analysis 3: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to the Inattention subscale score; Test type: Superiority; p = 0.0424, ANCOVA; Least Square Mean Difference = -2.1, 95% CI 2-sided [-4.2 to -0.1], Standard Error of Mean 1.05
Statistical Analysis 4: Comparison: Placebo vs 400mg SPN-812; This analysis pertains to the Inattention subscale score; Test type: Superiority; p = 0.0390, ANCOVA; Least Square Mean Difference = -2.1, 95% CI 2-sided [-4.1 to -0.1], Standard Error of Mean 1.03

8. Secondary Outcome: Effect of SPN-812 Assessed by Conners 3rd Edition - Self Report Short Form (C3-SRS)
Description: An additional secondary endpoint was the change from baseline in the Conners 3rd Edition - Self Report Short Form (C3-SRS) Composite T score at Week 6 (End of Study). The Conners 3rd Edition is a focused diagnostic tool for assessment of ADHD and associated learning, behavior, and emotional problems in children 6 to 18 years of age. The C3-SRS, which is only validated in children/adolescents 8-18 years of age, is comprised of 41 items with subsets of items related to five content scales: inattention, hyperactivity/impulsivity, learning problems, aggression and family relations. The subject rates himself/herself on the first 39 items of C3-SRS using a 4-point Likert scale (0-3; where 0=not at all true [never, seldom] and 3=very much true [very often, very frequently] based on past month; the last 2 items are fill-in-the-blank and do not contribute to the raw score(s). Raw scores are converted to T-scores. Lower change from baseline T-scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 104 | 94 | 103
T-score | -4.4 (0.82) | -5.5 (0.88) | -4.5 (0.83)
Statistical Analysis 1: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.3813, ANCOVA; Least Square Mean Difference = -1.0, 95% CI 2-sided [-3.4 to 1.3], Standard Error of Mean 1.20
Statistical Analysis 2: Comparison: Placebo vs 400mg SPN-812; Test type: Superiority; p = 0.9506, ANCOVA; Least Square Mean Difference = -0.1, 95% CI 2-sided [-2.4 to 2.2], Standard Error of Mean 1.17

9. Secondary Outcome: Effect of SPN-812 Assessed by Categorical Clinical Global Impression - Improvement (CGI-I) [the Percentage of Subjects Who Were 'Improved"]
Description: An additional secondary endpoint was the percentage of subjects who were "improved" by visit; "improved" was defined as a subject who had a Clinical Global Impression - Improvement (CGI-I) score of 1 = "Very Much Improved" or 2 = "Much Improved". Values range from 0 to 100%. A higher percentage represents a greater number of subjects who were "improved".
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 104 | 94 | 103
percentage of subjects
  Week 1 | 4.8 | 14.1 | 16.5
  Week 2 | 17.0 | 27.0 | 32.1
  Week 3 | 21.9 | 39.8 | 46.3
  Week 4 | 28.5 | 49.4 | 55.6
  Week 5 | 32.5 | 51.9 | 53.7
  Week 6 | 31.6 | 50.7 | 51.9
Statistical Analysis 1: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 1; Test type: Superiority; p = 0.0254, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 2; Test type: Superiority; p = 0.0899, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 3; Test type: Superiority; p = 0.0070, Chi-squared
Statistical Analysis 4: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 4; Test type: Superiority; p = 0.0031, Chi-squared
Statistical Analysis 5: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 5; Test type: Superiority; p = 0.0065, Chi-squared
Statistical Analysis 6: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 6; Test type: Superiority; p = 0.0070, Chi-squared
Statistical Analysis 7: Comparison: Placebo vs 400mg SPN-812; This analysis pertains to Week 1; Test type: Superiority; p = 0.0063, Chi-squared
Statistical Analysis 8: Comparison: Placebo vs 400mg SPN-812; This analysis pertains to Week 2; Test type: Superiority; p = 0.0123, Chi-squared
Statistical Analysis 9: Comparison: Placebo vs 400mg SPN-812; This analysis pertains to Week 3; Test type: Superiority; p = 0.0003, Chi-squared
Statistical Analysis 10: Comparison: Placebo vs 400mg SPN-812; This analysis pertains to Week 4; Test type: Superiority; p = 0.0001, Chi-squared
Statistical Analysis 11: Comparison: Placebo vs 400mg SPN-812; This analysis pertains to Week 5; Test type: Superiority; p = 0.0025, Chi-squared
Statistical Analysis 12: Comparison: Placebo vs 400mg SPN-812; This analysis pertains to Week 6; Test type: Superiority; p = 0.0033, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The number of subjects reported in each arm for Adverse Events table is based on the Safety Population (actual treatment arm); includes subjects who were randomized and took at least one dose of study medication. One subject was randomized to the 400mg SPN-812 arm (assigned treatment arm), but received 200mg SPN-812 during the trial (actual treatment arm). Therefore, the number of participants between SPN-812 arms will differ by 1 between the Participant Flow table and Adverse Events table.
Arm/Group | Placebo | 200mg SPN-812 | 400mg SPN-812
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/99 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/104 | 2/99 | 0/105
Other Adverse Events (participants affected / at risk) | 22/104 | 39/99 | 50/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=104) | 200mg SPN-812 (N=99) | 400mg SPN-812 (N=105)
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=104) | 200mg SPN-812 (N=99) | 400mg SPN-812 (N=105)
Somnolence (Nervous system disorders) | 8 | 13 | 15
Headache (Nervous system disorders) | 10 | 10 | 13
Decreased appetite (Metabolism and nutrition disorders) | 0 | 5 | 9
Nausea (Gastrointestinal disorders) | 3 | 7 | 7
Fatigue (General disorders) | 1 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03247517/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03247517/SAP_001.pdf